CLINICAL TRIAL: NCT05840302
Title: Effectiveness of a Pain Neuroscience Education Programme on Physical Activity in Patients With Chronic Low Back Pain. Randomised Controlled Trial
Brief Title: Effectiveness of a Pain Neuroscience Education Programme on Physical Activity in Patients With Chronic Low Back Pain
Acronym: END-LC
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Montpellier (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: RECHMPL21_0513; ID-RCB (Registry Identifier: 2023-A00346-39)
Record Dates: First submitted 2023-04-21; First posted 2023-05-03 (Actual); Last update posted 2025-09-30 (Actual); Status verified 2025-09

CONDITIONS: Low Back Pain, Recurrent
Keywords: Low back pain; Pain Neurosciences Education; Physical activity
MeSH Terms: conditions — Low Back Pain; Motor Activity | interventions — Fitness Trackers; Surveys and Questionnaires

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Pain Neuroscience Education (Experimental): The Pain Neuroscience Education program takes place over ten days consisting of providing knowledge about the neurophysiology and central processes of pain (nociceptive pathways, inhibitory circuits, peripheral and central sensitization, nervous system plasticity) as well as psychosocial factors and beliefs contributing to chronic pain. Workshops will use experimental data from neuroscience, but also analogies, brainstorming or games. Questions are proposed to the patient at the end of each theme.
  Interventions: Device: Activity monitor; Other: Questionnaire
- Back School (Active Comparator): The Back School program takes place over ten days. It begins with a presentation of spinal economy, which consists of promoting the protection of the back. Then, the anatomy and biomechanics of the spine as well as the most common spinal pathologies are presented. On this biomechanical basis, the other sessions consist in indicating the gestures and postures to adopt, always according to the protection policy, in different situations. These different sessions alternate between theory and practical exercises.
  Interventions: Device: Activity monitor; Other: Questionnaire

INTERVENTIONS:
Device: Activity monitor — Measure of number of steps and physical activity during one week using the activity monitor (connected watch) named the ActiGraph-wGT3X-BT medical device, Pre-test before intervention, post-test 3-months and 1-year after intervention
Other: Questionnaire — Self and hetero assessments measuring pain, different determinants of chronic pain and physical activity

SUMMARY:
Proposing ways to effectively counter chronic low back pain through non-drug intervention is a major public health issue due to the prevalence and health costs of this condition. The back school (BS) is based on spinal economics and a biomechanical model. A convergence of evidence indicates that this type of program does not bring any mid- or long-term benefit. Faced with this observation, a Pain Neuroscience Education (PNE) has been developed based on a biopsychosocial model. Chronic low back pain is the consequence of a complex dynamic of multifactorial origin where the body lesion is no longer the only cause of the pain. Studies have shown that PNE has a positive effect on pain perception. One of the limitations of these studies is that they do not allow objective measurement of physical activity performed at a distance from a therapeutic program for patients who have benefited from these educational programs. Yet, physical activity is an essential variable in health and more specifically in the fight against pain in patients with chronic low back pain.

The investigators believe that physical activity is a key factor in improving the condition of patients with chronic low back pain. Consequently, physical activity is an indicator of success but also a guarantee for a lasting effect of educational treatment. In order to measure this physical activity, the use of activity monitor (connected watch) developed in recent years now makes it possible to collect data in an ecological manner that is more objective than the data collected via self-questionnaires.

The main objective of the study is to measure the effectiveness of a PNE on physical activity three months after the intervention compared to BS in patients with chronic low back pain receiving a multidisciplinary rehabilitation program.

The secondary aims are to compare effectiveness of PNE versus BS on pain, quality of life, kinesiophobia, pain catastrophizing, central sensitization at 3 months and at one year after the intervention. In addition, an exploratory analysis will be conducted to determine predictors of physical activity maintenance.

The investigators expect to observe greater physical activity in patients who have received a PNE program compared to the physical activity of patients who have completed an BS program.

ELIGIBILITY:
Inclusion Criteria:

* Patient over 18 years of age.
* Ordinary back pain according to the High Authority for Health criteria 2019
* Chronic back pain (> 3months)
* Start Back Screening Tool > 3
* Partial hospitalization at the Lamalou-les-Bains Hospital for a multidisciplinary rehabilitation program

Exclusion Criteria:

* Subject with a comorbidity that limits walking (e.g. central neurological disorder)
* Subject with current psychiatric or cognitive co-morbidity that does not allow educational programs to be completed
* Stay following a surgical procedure of less than three months
* Other specific low back pain treatment planned during the 3 months of follow-up (surgery, infiltration)
* Patient participating in another clinical trial related to low back pain
* Subject does not understand the French language.
* Pregnant woman, parturient or nursing
* Subject with a legal protection measure (guardianship, curators)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 82 (Estimated)
Dates: Start 2023-10-02 (Actual); Primary Completion 2027-09 (Estimated); Study Completion 2027-09 (Estimated)

PRIMARY OUTCOMES:
Number of Steps 3 months after rehabilitation program | 3 months after rehabilitation program
  Comparison between the two arms of the average number of daily steps calculated over 7 days by an activity monitor (connected watch) named Actigraph wGT3X-BT

SECONDARY OUTCOMES:
Changes in Number of Steps 3 months after rehabilitation program | between baseline and 3 months
  Changes in the average number of daily steps calculated over 7 days by an activity monitor (connected watch) named Actigraph wGT3X-BT at two different times (before and 3 months after rehabilitation program)
Changes in Number of Steps 12 months after rehabilitation program | between 3 months and 12 months
  Changes in the average number of daily steps calculated over 7 days by an activity monitor (connected watch) named Actigraph wGT3X-BT at two different times (3 and 12 months after rehabilitation program)
Number of Steps 12 months after rehabilitation program | 12 months after rehabilitation program
  Comparison between the two arms of the average number of daily steps calculated over 7 days by an an activity monitor (connected watch) named Actigraph wGT3X-BT
Pain intensity 3 months after rehabilitation program | 3 months after rehabilitation program
  Comparison between the two arms of the pain intensity. Pain intensity score will evaluated using a Pain Numerical Rating Scale (NRS) A high score indicates severe pain (0 = absence of pain, 10 = severe pain)
Pain intensity 12 months after rehabilitation program | 12 months after rehabilitation program
  Comparison between the two arms of the pain intensity. Pain intensity score will evaluated using a Pain Numerical Rating Scale (NRS) A high score indicates severe pain (0 = absence of pain, 10 = severe pain)
Changes in pain intensity 3 months after rehabilitation program | between baseline and 3 months
  Changes in pain intensity at two different times (before and 3 months after rehabilitation program) Pain intensity score will evaluated using a Pain Numerical Rating Scale (NRS) A high score indicates severe pain (0 = absence of pain, 10 = severe pain)
Changes in pain intensity 12 months after rehabilitation program | between 3 and 12 months
  Changes in pain intensity at two different times (before and 3 months after rehabilitation program) Pain intensity score will evaluated using a Pain Numerical Rating Scale (NRS) A high score indicates severe pain (0 = absence of pain, 10 = severe pain)
Central Sensitivity score 3 months after rehabilitation program | 3 months after rehabilitation program
  Comparison between the two arms of the Central Sensitivity score Central Sensitivity score will evaluate with The Central Sensitization Inventory that is a valid screening tool to identify and quantify central sensitization to pain
Central Sensitivity score 12 months after rehabilitation program | 12 months after rehabilitation program
  Comparison between the two arms of the Central Sensitivity score Central Sensitivity score will evaluate with The Central Sensitization Inventory that is a valid screening tool to identify and quantify central sensitization to pain
Changes in Central Sensitivity score 3 months after rehabilitation program | between baseline and 3 months
  Changes in Central Sensitivity score at two different times (before and 3 months after rehabilitation program). Central Sensitivity score will evaluate with The Central Sensitization Inventory that is a valid screening tool to identify and quantify central sensitization to pain
Changes in Central Sensitivity score 12 months after rehabilitation program | between 3 and 12 months
  Changes in pain intensity at two different times (3 and 12 months after rehabilitation program). Central Sensitivity score will evaluate with The Central Sensitization Inventory that is a valid screening tool to identify and quantify central sensitization to pain
Pain Catastrophizing score 3 months after rehabilitation program | 3 months after rehabilitation program
  Comparison between the two arms of the Pain Catastrophizing score. The Pain Catastrophizing Scale is a questionnaire of 13 statements rated by a five-point ordinal scale, measuring a subject's level of pain catastrophizing.
Pain Catastrophizing score 12 months after rehabilitation program | 12 months after rehabilitation program
  Comparison between the two arms of the Pain Catastrophizing score. The Pain Catastrophizing Scale is a questionnaire of 13 statements rated by a five-point ordinal scale, measuring a subject's level of pain catastrophizing.
Changes in Pain Catastrophizing score 3 months after rehabilitation program | between baseline and 3 months
  Changes in the Pain Catastrophizing score at two different times (baseline and 3 months after rehabilitation program) The Pain Catastrophizing Scale is a questionnaire of 13 statements rated by a five-point ordinal scale, measuring a subject's level of pain catastrophizing.
Changes in Pain Catastrophizing score 12 months after rehabilitation program | between 3 and 12 months
  Changes in the Pain Catastrophizing score at two different times (3 and 12 months after rehabilitation program) The Pain Catastrophizing Scale is a questionnaire of 13 statements rated by a five-point ordinal scale, measuring a subject's level of pain catastrophizing.
Kinesiophobia scale score 3 months after rehabilitation program | 3 months after rehabilitation program
  Comparison between the two arms of the Kinesiophobia scale score Kinesiophobia scale score will evaluate using the Tampa Scale of Kinesiophobia. The Tampa Scale of Kinesiophobia is a questionnaire of 17 questions rated by a four-point ordinal scale, measuring the fear that pain may occur as a result of movement. These fears can lead to avoidance behaviors and reduced activity
Kinesiophobia scale score 12 months after rehabilitation program | 12 months after rehabilitation program
  Comparison between the two arms of the Kinesiophobia scale score Kinesiophobia scale score will evaluate using the Tampa Scale of Kinesiophobia. The Tampa Scale of Kinesiophobia is a questionnaire of 17 questions rated by a four-point ordinal scale, measuring the fear that pain may occur as a result of movement. These fears can lead to avoidance behaviors and reduced activity
Changes in Kinesiophobia scale score 3 months after rehabilitation program | between baseline and 3 months
  Changes in the Pain Catastrophizing score at two different times (baseline and 3 months after rehabilitation program) Kinesiophobia scale score will evaluate using the Tampa Scale of Kinesiophobia. The Tampa Scale of Kinesiophobia is a questionnaire of 17 questions rated by a four-point ordinal scale, measuring the fear that pain may occur as a result of movement. These fears can lead to avoidance behaviors and reduced activity
Changes in Kinesiophobia scale score 12 months after rehabilitation program | between 3 and 12 months
  Changes in the Pain Catastrophizing score at two different times (3 and 12 months after rehabilitation program) Kinesiophobia scale score will evaluate using the Tampa Scale of Kinesiophobia. The Tampa Scale of Kinesiophobia is a questionnaire of 17 questions rated by a four-point ordinal scale, measuring the fear that pain may occur as a result of movement. These fears can lead to avoidance behaviors and reduced activity
Canadian Occupational Performance Measure 3 months after rehabilitation program | 3 months after rehabilitation program
  Comparison between the two arms of Canadian Occupational Performance Measure The Canadian Occupational Performance Measure assess changes in occupational during a semi-structured interview performance
Canadian Occupational Performance Measure 12 months after rehabilitation program | 12 months after rehabilitation program
  Comparison between the two arms of Canadian Occupational Performance Measure The Canadian Occupational Performance Measure assess changes in occupational during a semi-structured interview performance
Changes in Canadian Occupational Performance Measure 3 months after rehabilitation program | between baseline and 3 months
  Changes in the Pain Catastrophizing score at two different times (baseline and 3 months after rehabilitation program). The Canadian Occupational Performance Measure assess changes in occupational during a semi-structured interview performance.
Changes in Canadian Occupational Performance Measure 12 months after rehabilitation program | between 3 and 12 months
  Changes in the Pain Catastrophizing score at two different times (3 and 12 months after rehabilitation program). The Canadian Occupational Performance Measure assess changes in occupational during a semi-structured interview performance.
Global Physical Activity score 3 months after rehabilitation program | 3 months after rehabilitation program
  Comparison between the two arms of the Global Physical Activity score. Global Physical Activity score will evaluate using the Global Physical Activity Questionnaire.
  The Global Physical Activity Questionnaire consists of 16 questions designed to estimate an individual's level of physical activity in 3 domains (work, transport and leisure time) and time spent in sedentary behavior
Global Physical Activity score 12 months after rehabilitation program | 12 months after rehabilitation program
  Comparison between the two arms of the Global Physical Activity score. Global Physical Activity score will evaluate using the Global Physical Activity Questionnaire.
  The Global Physical Activity Questionnaire consists of 16 questions designed to estimate an individual's level of physical activity in 3 domains (work, transport and leisure time) and time spent in sedentary behavior
Changes in the global Physical Activity score 3 months after rehabilitation program | between baseline and 3 months
  Changes in the global Physical Activity score at two different times (baseline and 3 months after rehabilitation program). Global Physical Activity score will evaluate using the Global Physical Activity Questionnaire.
  The Global Physical Activity Questionnaire consists of 16 questions designed to estimate an individual's level of physical activity in 3 domains (work, transport and leisure time) and time spent in sedentary behavior
Changes in the global Physical Activity score 12 months after rehabilitation program | between 3 and 12 months
  Changes in the global Physical Activity score at two different times (3 and 12 months after rehabilitation program). Global Physical Activity score will evaluate using the Global Physical Activity Questionnaire.
  The Global Physical Activity Questionnaire consists of 16 questions designed to estimate an individual's level of physical activity in 3 domains (work, transport and leisure time) and time spent in sedentary behavior
Hospital Anxiety and Depression score 3 months after rehabilitation program | 3 months after rehabilitation program
  Comparison between the two arms of the Hospital Anxiety and Depression score Hospital Anxiety and Depression score will evaluate using Hospital Anxiety and Depression scale.
  The Hospital Anxiety and Depression Scale consists of 7 items designed to evaluate depression and 7 for the anxiety.
Hospital Anxiety and Depression score 12 months after rehabilitation program | 12 months after rehabilitation program
  Comparison between the two arms of the Hospital Anxiety and Depression score Hospital Anxiety and Depression score will evaluate using Hospital Anxiety and Depression scale.
  The Hospital Anxiety and Depression Scale consists of 7 items designed to evaluate depression and 7 for the anxiety.
Changes in Hospital Anxiety and Depression score 3 months after rehabilitation program | between baseline and 3 months
  Changes in Hospital Anxiety and Depression score at two different times (baseline and 3 months after rehabilitation program).
  Hospital Anxiety and Depression score will evaluate using Hospital Anxiety and Depression scale.
  The Hospital Anxiety and Depression Scale consists of 7 items designed to evaluate depression and 7 for the anxiety.
Changes in Hospital Anxiety and Depression score 12 months after rehabilitation program | between baseline and 12 months
  Changes in Hospital Anxiety and Depression score at two different times (3 and 12 months after rehabilitation program).
  Hospital Anxiety and Depression score will evaluate using Hospital Anxiety and Depression scale.
  The Hospital Anxiety and Depression Scale consists of 7 items designed to evaluate depression and 7 for the anxiety.
Quality of Life Score 3 months after rehabilitation program | 3 months after rehabilitation program
  Comparison between the two arms of the Quality of Life Score The Quality of Life Score will evaluate with the Short Form (36) Health Survey questionnaire that is multidimensional assessment of quality of life
Quality of Life Score 12 months after rehabilitation program | 12 months after rehabilitation program
  Comparison between the two arms of the Quality of Life Score The Quality of Life Score will evaluate with the Short Form (36) Health Survey questionnaire that is multidimensional assessment of quality of life
Changes in the Quality of Life Score 3 months after rehabilitation program | between baseline and 3 months after rehabilitation
  Changes in Quality of Life Score at two different times (baseline and 3 months after rehabilitation program).
  The Quality of Life Score will evaluate with the Short Form (36) Health Survey questionnaire that is multidimensional assessment of quality of life
Changes in the Quality of Life Score 12 months after rehabilitation program | between 3 and 12 months after rehabilitation program
  Changes in Quality of Life Score at two different times (3 and 12 months after rehabilitation program). The Quality of Life Score will evaluate with the Short Form (36) Health Survey questionnaire that is multidimensional assessment of quality of life

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital Center Paul Coste Floret, Lamalou-les-Bains, France

REFERENCES:
- [Derived] Thebault G, Duflos C, Le Perf G. Effectiveness of a pain neuroscience education programme on the physical activity of patients with chronic low back pain compared with a standard back school programme: protocol for a randomised controlled study (END-LC). BMJ Open. 2024 Jun 3;14(6):e080079. doi: 10.1136/bmjopen-2023-080079. PMID 38830744